CLINICAL TRIAL: NCT06956066
Title: THE EFFECT OF SUBCUTANEOUS "SHOTBLOCKER" ON INJECTION PAIN, ANXIETY AND COMFORT LEVEL IN GERIATRIC PATIENTS
Brief Title: The Effect of SHOTBLOCKER
Acronym: SHOTBLOCKER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Berna Dincer, Nursing Associate Professor, Istanbul Medeniyet University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IstanbulMU
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Shotblocker; Injection Pain Prevention; Pain; Anxiety
Keywords: Shotblocker; injection; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Assuming a power of 80% and an α risk of. 05, a sample size of 75 was determined to be appropriate. Considering the possibility of missing data, the study initially included 80 participants in both the experimental and control groups. A computer-based random number generator was used for group assignment, and allocation concealment was ensured by using sealed envelopes containing random numbers opened by a separate researcher. The study was completed with 40 participants in the experimental group and 40 in the control group, due to some participants withdrawing.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shotblocker (Experimental): injection with shotblocker
  Interventions: Biological: shotblocker
- Control (No Intervention): Normal injection

INTERVENTIONS:
Biological: shotblocker — SHOTBLOCKER Shotblocker is a drug-free and non-invasive plastic device for all age groups that is placed during injection to press against the site of administration. It has standardized dimensions and is designed in a small, flat, horseshoe (U) shape with several blunt points on one surface in direct contact with the skin.
  Arms: shotblocker

SUMMARY:
This study was conducted as a randomized controlled experimental cross over study to examine the effect of injection pain, anxiety and comfort level with the use of Shotblocker in geriatric patients undergoing subcutaneous injection. The study was defined on 80 patients who were inpatients in the internal wards of a hospital, and the experimental and control groups, which provided the appropriate conditions for the study, included the same people. Ethics committee approval, institutional permission and written informed consent forms were obtained from the individuals. Data were obtained by the researcher using Personal Information Form, Visual Analog Scale (VAS), State and Trait Anxiety Scale, Comfort Scale, Visual Patient Satisfaction Scale and Shotblocker.

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled experimental cross over study to examine the effect of injection pain, anxiety and comfort level with the use of Shotblocker in geriatric patients undergoing subcutaneous injection. The study was defined on 80 patients who were inpatients in the internal wards of a hospital, and the experimental and control groups, which provided the appropriate conditions for the study, included the same people. Ethics committee approval, institutional permission and written informed consent forms were obtained from the individuals. Data were obtained by the researcher using Personal Information Form, Visual Analog Scale (VAS), State and Trait Anxiety Scale, Comfort Scale, Visual Patient Satisfaction Scale and Shotblocker.

ELIGIBILITY:
Inclusion Criteria:

Voluntary participants in the study, Over 65 years of age, Cognitive ability to answer the questions, Body Mass Index (BMI) 18.5- 29.9 kg / m2, No communication problems, Subcutaneous injection in the treatment, No bleeding coagulation disorder, Platelet, INR and APTT values within normal limits, No scar tissue, incision or infection findings in the injection area, No history of allergy

Exclusion Criteria:

Patients with amputation in the right/left arm area to be studied, Patients with any scar tissue, incision, lipodystrophy or signs of infection in the injection area in the arm area, Patients receiving hemodialysis treatment and having a dialysis catheter, Patients who underwent mastectomy surgery and should not undergo any application/treatment on the arm on the operated side were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory | Time Frame: up to 1 day
  1. Beck Anxiety Inventory Description: It is a Likert-type scale consisting of 21 items and scored between 0-3. According to scale scoring; 8 points: No anxiety, 8-15 points: Mild anxiety, 16-25 points: Moderate anxiety, 26-63 points: Determined as severe anxiety decrease the15 points

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No